CLINICAL TRIAL: NCT02002832
Title: A Randomized, Double-blind, Double-dummy, Parallel-group and Multicenter Study to Investigate Lurasidone in Treatment of Schizophrenia Compared With Risperidone
Brief Title: A Clinical Trial of Lurasidone in Treatment of Schizophrenia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sumitomo Pharma (Suzhou) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D1070004
Record Dates: First submitted 2013-12-02; First posted 2013-12-06 (Estimated); Results first posted 2019-04-01 (Actual); Last update posted 2019-11-15 (Actual); Status verified 2018-05

CONDITIONS: Schizophrenia
Keywords: schizophrenia; Lurasidone; LATUDA
MeSH Terms: conditions — Schizophrenia | interventions — Lurasidone Hydrochloride; Risperidone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lurasidone group (Experimental)
  Interventions: Drug: Lurasidone tablets
- Risperidone group (Active Comparator)
  Interventions: Drug: Risperidone tablets

INTERVENTIONS:
Drug: Lurasidone tablets — Lurasidone tablets (40or80mg/day) and Risperidone tablets(Placebo)
  Other Names: LATUDA
  Arms: Lurasidone group
Drug: Risperidone tablets — Risperidone tablets(2-6mg/day) and Lurasidone tablets(Placebo)
  Arms: Risperidone group

SUMMARY:
This is a randomized, double-blind, double-dummy, parallel- controlled, adjustable dose, non-inferiority and multicentre study designed to evaluate the efficacy and safety of lurasidone on schizophrenia for 6 weeks treatment, and to compare with risperidone.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent and aged between 18 and 65 years of age.
* Meets DSM-IV-TR criteria for a primary diagnosis of schizophrenia, had a PANSS total score ≥ 70 and ≤ 120 at Screening and Baseline, and a score ≥ 4 on the CGI-S at Screening and Baseline.
* Not pregnant, if of reproductive potential agrees to use adequate and reliable contraception for duration of study.
* Able and agrees to remain off prior antipsychotic medication for the duration of study.
* Willing and able to comply with the protocol, including the inpatient requirements and outpatient visits.

Exclusion Criteria:

* Considered by the investigator to be at imminent risk of suicide or injury to self, others or property.
* Any chronic organic disease of the CNS(other than schizophrenia)
* Subjects are participating or participated in other clinical studies including marketed drugs or medical devices within 30 days before signing the informed consent form.
* Clinically significant or history of alcohol abuse/alcoholism or drug abuse/dependence within the last 6 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 388 (Actual)
Dates: Start 2013-12; Primary Completion 2015-04 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zhuoji CAI, MD, Principal Investigator — Capital Medical University Affiliated Beijing Anding Hospital
Locations (15):
- China (15):
  - Capital Medical University Affiliated Beijing Anding Hospital, Beijing, Beijing Municipality
  - Beijing Huilongguan Hospital, Beijing, Beijing Municipality
  - Peking University Sixth Hospital, Beijing, Beijing Municipality
  - Guangzhou Brain Hospital, Guangzhou, Guangdong
  - HeBei Mental Health Center, Baoding, Hebei
  - Henan Provincial Mental Hospital, Xinxiang, Henan
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - Hunan Province Brain Hospital, Changsha, Hunan
  - Nanjing Brain Hospital, Nanjing, Jiangsu
  - Wuxi Mental Health Center, Wuxi, Jiangsu
  - Shanghai Mental Health Center, Shanghai, Shanghai Municipality
  - Xi'an Mental Health Center, Xi’an, Shanxi
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Tianjin Anding Hospital, Tianjin, Tianjin Municipality
  - First Affiliated Hospital of Kunming Medical University, Kunming, Yunnan

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Lurasidone Group: Lurasidone 40 or 80 mg tablets taken orally once a day and Risperidone placebo tablets taken orally once a day
- Risperidone Group: Risperidone 2-6mg tablets taken orally once a day and Lurasidone placebo tablets taken orally once a day.
Period: Overall Study
Arm/Group | Lurasidone Group | Risperidone Group
Started | 194 | 194
Completed | 166 | 168
Not Completed | 28 | 26

BASELINE CHARACTERISTICS:
Population: Intent-to-treat population (ITT) : All randomized subjects who received at least one dose of study medication,were included in the Intent-to-treat population.
Groups:
- Risperidone Group: Risperidone 2-6mg taken orally once a day and Lurasidone placebo tablets taken orally once a day.
- Total: Total of all reporting groups
Arm/Group | Lurasidone Group | Risperidone Group | Total
Number analyzed (Participants) | 194 | 190 | 384
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 194 | 190 | 384
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.6 (11.12) | 34.8 (10.71) | 34.7 (10.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 96 | 89 | 185
  Male | 98 | 101 | 199
Region of Enrollment [Number; unit: participants]
  China | 194 | 190 | 384

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline to Week 6 in Positive and Negative Syndrome Scale (PANSS) Total Scores.
Description: Mean change in Positive and Negative Syndrome Scale total score from baseline to Week 6 at the end of treatment. PANSS is an interview-based measure of the severity of psychopathology in adults with psychotic disorders. It have 30 evaluation items, which include 7 positive sub-scale, 7 negative sub-scale and 16 general psychopathology sub-scale on a score of 1 to 7. The total score is the sum of the 30 scale items. The minimum score is 30 and the maximum score is 210. Patient with PANSS total scores<70 is the normal,but the scores>120 is more serious.
Time Frame: From baseline to Week 6(day 42).
Population: Intent-to-Treat population: All subjects who were randomized, received at least one dose of study medication, and have a Baseline efficacy measurement and at least one post-Baseline efficacy measurement, were in the efficacy analysis in the treatment group to which they were randomized.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Lurasidone Group | Risperidone Group
Number analyzed (Participants) | 194 | 190
units on a scale | -31.2 [-33.2 to -29.2] | -34.9 [-36.8 to -32.9]
Statistical Analysis 1: Comparison: Lurasidone Group vs Risperidone Group; Test type: Non-Inferiority or Equivalence — LS mean for the treatment difference(lurasidone-risperidone) at week 6 and its 95% confidence interval was presented based on the MMRM. Non-inferiority for lurasidone relative to risperidone was evaluated by comparing the upper bound of the 95% confidence interval to the non-inferiority margin of 7.0. Plots of estimates for change from baseline in PANSS total score based on MMRM over time (Week 1 to Week 6) with 95% confidence intervals was provided for each treatment group; Mixed Models Analysis; Mean Difference (Final Values) = 3.7, 95% CI 2-sided [1.0 to 6.3], Standard Error of Mean 1.37

2. Secondary Outcome: Mean Clinical Global Impression Scale-Improvement (CGI-I) Score at Week 6.
Description: The Clinical Global Impression Scale-Improvement (CGI-I) Score is a 7 point scale that requires the clinician to assess how much the patient's illness has improved or worsened relative to baseline state at the beginning of the intervention. Response is rated as one of the following, in which higher scores indicate less improvement or worsening:
  1=Very much improved, 2=Much improved, 3=Minimally improved, 4=No change, 5=Minimally worse, 6=Much worse, and 7=Very much worse.
Time Frame: From baseline to Week 6(day 42).
Population: The primary population for the efficacy analysis was the Intent-to-Treat (ITT) population. All subjects who were randomized, received at least one dose of study medication, and have a Baseline efficacy measurement and at least one post-Baseline efficacy measurement, were in the efficacy analysis in the treatment group to which they were randomized.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Lurasidone Group | Risperidone Group
Number analyzed (Participants) | 194 | 190
units on a scale | 2.0 [1.9 to 2.1] | 1.9 [1.8 to 2.0]

ADVERSE EVENTS:
Time Frame: Date of first dose of study medication and up to 7 days after date of last dose of treatment in double-blind phase, an average of 7 weeks.
Description: Of the 388 randomized subjects, 385 subjects received at least 1 dose of study medication and were therefore included in the Safety population: 194 (100%) in the lurasidone group and 191 (98.5%) in the risperidone group.
Arm/Group | Lurasidone Group | Risperidone Group
All-Cause Mortality (participants affected / at risk) | 0/194 | 0/191
Serious Adverse Events (participants affected / at risk) | 1/194 | 0/191
Other Adverse Events (participants affected / at risk) | 134/194 | 160/191
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lurasidone Group (N=194) | Risperidone Group (N=191)
Hand fracture (Injury, poisoning and procedural complications) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lurasidone Group (N=194) | Risperidone Group (N=191)
Extrapyramidal disorder (Nervous system disorders) | 33 | 73
Akathisia (Nervous system disorders) | 14 | 26
Dizziness (Nervous system disorders) | 5 | 8
Poor quality sleep (Nervous system disorders) | 3 | 7
Hypertonia (Nervous system disorders) | 2 | 6
Consitpation (Gastrointestinal disorders) | 25 | 28
Nausea (Gastrointestinal disorders) | 7 | 4
Vomiting (Gastrointestinal disorders) | 6 | 3
Diarrhoea (Gastrointestinal disorders) | 5 | 5
Insomnia (Psychiatric disorders) | 19 | 19
Anxiety (Psychiatric disorders) | 12 | 12
Initial insomnia (Psychiatric disorders) | 7 | 6
Agitation (Psychiatric disorders) | 5 | 3
Affect lability (Psychiatric disorders) | 4 | 1
Nasopharyngitis (Infections and infestations) | 19 | 28
Upper respiratory tract infection (Infections and infestations) | 10 | 16
Hepatic function abnormal (Hepatobiliary disorders) | 8 | 6
Sinus bradycardia (Cardiac disorders) | 7 | 4
Sinus tachycardia (Cardiac disorders) | 2 | 7
Tachycardia (Cardiac disorders) | 1 | 5
Blood prolactin increased (Investigations) | 6 | 27
Transaminases increased (Investigations) | 2 | 6
Weight increased (Investigations) | 1 | 10
Asthenia (General disorders) | 3 | 5
Anaemia (Blood and lymphatic system disorders) | 2 | 4
Vision blurred (Eye disorders) | 1 | 4
Decreased appetite (Metabolism and nutrition disorders) | 1 | 4
Hyperprolactinaemia (Endocrine disorders) | 1 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No